CLINICAL TRIAL: NCT02428738
Title: Text Message Reminders for Influenza Vaccine in Pregnancy
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 13-265
Record Dates: First submitted 2015-04-16; First posted 2015-04-29 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy
Keywords: Influenza Vaccine; Text Message
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Influenza virus accounts for numerous cases (epidemics) of respiratory illnesses each year worldwide and affects people of all ages. These epidemics typically occur in the winter months, and can result in substantial morbidity and mortality in persons at risk. Pregnant women may be more susceptible to morbidity and mortality associated with influenza infection. This increased risk may result from several factors including increased heart rate, stroke volume, and oxygen consumption, decreased lung capacity, and changes in immunologic function. Immunization of women during pregnancy can help to prevent infection in the woman herself and may also offer protection to the infant in two ways: by the passage of antibodies from mother to the fetus during pregnancy, and by preventing infection in the mother and therefore decreasing the infant's exposure risk after birth. In Canada, the National Advisory Committee on Immunization (NACI) recommends the vaccine for pregnant women who are expected to deliver during influenza season because they will become household contacts of their newborn. Ideal timing of vaccination occurs in October or November since influenza outbreaks typically occur throughout the winter months. Despite the Canadian and American guidelines for influenza vaccination during pregnancy, it is unclear how many women are offered and/or actually receive the vaccine while pregnant. There is, however, evidence that women will accept the vaccine if offered. Specifically, in the Women's Health Care Centre at St. Michael's Hospital, it was found that 42% of women not only accepted but also received the influenza vaccination when offered. Innovative techniques will be required to continue to increase vaccination rates among vulnerable populations, including pregnant women. The purpose of the present study is to determine if the use of electronic reminders (text messages) increases the likelihood of receiving the influenza vaccine among pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Woman
* Ages 18 and over
* Working cellular telephone with the ability to receive text messages
* Ability to speak or understand English

Exclusion Criteria:

* Age less than 18
* Inability to speak or understand English
* Not possessing a working cellular telephone with text messaging capability
* Presence of any contraindications to vaccination (such as egg allergy or prior adverse reaction to the vaccine)
* Women who have already received the vaccine during this influenza season

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Women cared for in the Women's Health Care Centre prenatal clinic during influenza season
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of Influenza Vaccination of those who do receive text message reminders compared to those who do not. | Up to 5 months
  To determine the percentage of women who receive the influenza vaccine during pregnancy and also received text message reminders, relative to women who do not receive text messages.

SECONDARY OUTCOMES:
Patient characteristics affecting liklihood of receiving vaccine | Up to 5 months
  Patient characteristics (e.g. race/ethnicity, education level, family income, number of prior pregnancies, history of receiving the vaccine in the past) affecting the likelihood of receiving the vaccine among those who receive reminders.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yudin, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Yudin MH, Mistry N, De Souza LR, Besel K, Patel V, Blanco Mejia S, Bernick R, Ryan V, Urquia M, Beigi RH, Moniz MH, Sgro M. Text messages for influenza vaccination among pregnant women: A randomized controlled trial. Vaccine. 2017 Feb 1;35(5):842-848. doi: 10.1016/j.vaccine.2016.12.002. Epub 2017 Jan 3. PMID 28062124